CLINICAL TRIAL: NCT01753726
Title: Diaphragm Stretching Technique Increases Spine Mobility and Thoracic Movement: a Randomized Controlled Trial
Brief Title: Diaphragm Stretching Increases Spine and Thoracic Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DF0037UG
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: stretching, diaphragm, spinal movement, thoracic movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): 43 people are recruited in order to the inclusion criteria for the study. They are healthy people. A diaphragm stretching technique was employed in this experimental group.
  Interventions: Other: Diaphragm stretching.
- Placebo group (Placebo Comparator): 37 healthy people were recruited in order to the inclusion criteria.
  Interventions: Other: Placebo.

INTERVENTIONS:
Other: Diaphragm stretching. — A manual technique of diaphragm stretching during 7 minutes. The participants were situated in a seated position.
  Other Names: Manual technique
  Arms: Experimental group
Other: Placebo. — Disconnected ultrasound was used for the 7 min as sham treatment
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Physical therapists have traditionally included various forms of manual therapy among the therapeutic approaches to spinal pathologies. The aim of this study was to evaluate the effect of diaphragmatic stretching on spine and thoracic movement in healthy adults.

DETAILED DESCRIPTION:
Spinal pain is a well recognized condition associated with significant personal and community burdens. Recent studies estimated the prevalence between 6 and 22% in neck pain, from 4-72% in thoracic pain and from 1.0% to 58.1% in low back pain, which increases with age. During the last decades numerous researches have been conducted on stretching effects, evidencing an increased muscle control, flexibility and range of motion. The main purpose of this investigation is to examine the effects of diaphragm stretching in spine and thoracic mobility in healthy subjects in order to apply the results in a specifics pathologies in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age: between 18 and 65 years old.

Exclusion Criteria:

* Pathological subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of lumbar mobility | up to 2 months
  Schober test is a flexion trunk test to evaluate lumbar spine mobility. During this test, while the patient is in the standing position, marks are made in the midpoint between the posterior superior iliac spines (PSISs) and 10 cm superiorly to this point.

SECONDARY OUTCOMES:
Assessment of trunk mobility | baseline, 2 months
  In Finger to floor test, the subjects were stood on a stool and asked to flex the trunk forward in order to reach as far as possible with both hands, without blending their knees.
Cervical mobility | baseline, 2 months.
  A Baseline Bubble Inclinometer, Fabrication Enterprises Incorporated, New York. USA, was used to measure de active range of motion of the cervical spine. The measurements were performed in two planes of movement, lateral flexion (frontal plane) the right and left side; and flexion-extension (sagittal plane)
Abdominal and Thoracic Dimensions and Kinematics | baseline, 2 months.
  Abdominal and thoracic dimensions and kinematics measurements can be used as an evaluative method for diaphragmatic breathing excursion to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance as achieved by all expiratory and inspiratory muscles

CONTACTS AND LOCATIONS:
Overall Officials: M. Carmen Valenza, PH MD, Principal Investigator — Department of Physical Therapy. University of Granada.
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Alvarez FJ, Valenza MC, Torres-Sanchez I, Cabrera-Martos I, Rodriguez-Torres J, Castellote-Caballero Y. Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. Braz J Phys Ther. 2016 Jun 16;20(5):405-411. doi: 10.1590/bjpt-rbf.2014.0169. PMID 27333481
- See also: González-ÁlvarezFJ, ValenzaMC, Torres-SánchezI, Cabrera-MartosI, Rodríguez-TorresJ, CastelloteY.Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. BrazJPhysTher.2016 — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1413-35552016005008108&lng=en&nrm=iso&tlng=en